CLINICAL TRIAL: NCT00559546
Title: Montelukast as a Controller of Atopic Syndrome
Acronym: MONTAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HUS7/E5/07
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2007-11-16 (Estimated); Status verified 2007-11

CONDITIONS: Seasonal Allergic Rhinitis; Allergic Conjunctivitis; Atopic Eczema; Asthma
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Conjunctivitis, Allergic; Dermatitis, Atopic; Asthma | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 3 weeks of Montelukast and 3 weeks of placebo treatment
  Interventions: Drug: montelukast
- 2 (Active Comparator): 3 weeks of placebo and 3 weeks of montelukast treatment
  Interventions: Drug: montelukast

INTERVENTIONS:
Drug: montelukast — 10 mg montelukast tablet each evening for 3 weeks or placebo for 3 weeks in cross-over manner

SUMMARY:
The purpose of the study is to find out if montelukast can be used to treat the various symptoms of allergic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Wheal diameter at least 4 mm in skin-prick test for both birch and timothy
* Allergic symptoms in both upper airways (allergic rhinitis) and lower airways (asthma-like symptoms or diagnosed asthma) and at least one of the following:

  * Allergic conjunctivitis
  * Atopic eczema
  * Oral symptoms from vegetables or fruits by cross reactivity to birch
  * Urticaria in allergen exposure

Exclusion Criteria:

* Need for regular treatment with glucocorticoids
* Current smoking
* Other major disease or need for regular drug treatment
* Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2007-03; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Allergic symptoms | 3 weeks

SECONDARY OUTCOMES:
Need for antihistamines or inhaled beta-2-agonists to relieve symptoms | 3 weeks
Exhaled nitric oxide concentration | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tari Haahtela, Professor, Principal Investigator — Skin and Allergy Hospital, Helsinki University Hospital
Locations (1):
- Skin and Allergy Hospital, Helsinki University Hospital, Helsinki, Finland

REFERENCES:
- [Derived] Lehtimaki L, Petays T, Haahtela T. Montelukast is not effective in controlling allergic symptoms outside the airways: a randomised double-blind placebo-controlled crossover study. Int Arch Allergy Immunol. 2009;149(2):150-3. doi: 10.1159/000189198. Epub 2009 Jan 6. PMID 19127072